CLINICAL TRIAL: NCT07320339
Title: Standard vs. Routine Blood Pressure Measurement in Pregnancy: Effects of Position and Diurnal Variation
Brief Title: The Aim of the Study is to Examine the Variation in Blood Pressure Between an Optimal Measurement (According to Established Guidelines in the Literature - Per Guidelines) and a 'Common' Measurement (Used by Nursing Teams - Per Common Practice) Among Women of Reproductive Age With and Without Hyperte
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0111-25
Record Dates: First submitted 2025-11-16; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Blood Pressure Measurement in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- variation in blood pressure between an optimal measurement and a 'common' measurement (Experimental)
  Interventions: Procedure: blood pressure measurement

INTERVENTIONS:
Procedure: blood pressure measurement — examine the variation in blood pressure between an optimal measurement (according to established guidelines in the literature - per guidelines) and a 'common' measurement (used by nursing teams - per common practice) among women of reproductive age with and without hypertention

SUMMARY:
The aim of the study is to examine the variation in blood pressure between an optimal measurement (according to established guidelines in the literature - per guidelines) and a 'common' measurement (used by nursing teams - per common practice) among women of reproductive age with and without hyperte

DETAILED DESCRIPTION:
Accurate blood pressure measurement is a cornerstone of the diagnosis and management of hypertension. The latest Clinical Practice Guidelines (AHA2020- International Society of Hypertension Global) emphasize several important steps for accurate blood pressure measurement, including choosing the correct cuff size, resting for five minutes, sitting with support for the back, feet flat on the floor, and legs uncrossed, and proper arm positioning (i.e., positioning the midpoint of the cuff at heart level with the arm supported on a table or work surface). Sitting measurements are preferred because of the large amount of data linking blood pressure measurements in this position to health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40
* Informed consent to participate.

Exclusion Criteria:

* Inability to cooperate with BP measurement under optimal conditions
* Women with complex underlying disease that may bias the data (e.g. significant vasculopathy)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — • Women aged 18-40
Enrollment: 500 (Estimated)
Dates: Start 2025-08-24 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Mean difference in systolic blood pressure (mmHg) between guideline-based and routine clinical measurement | 1 year
  Mean difference in systolic blood pressure (mmHg) between guideline-based and routine clinical measurement
  Description:
  Systolic blood pressure (SBP) will be measured in each participant using two methods:
  1. guideline-based blood pressure measurement performed according to international hypertension guidelines (seated position, appropriate cuff size, arm supported at heart level after ≥5 minutes of rest), and
  2. routine clinical blood pressure measurement as performed by nursing staff under usual clinical conditions.
  The primary outcome will be the within-participant mean difference in SBP (mmHg) between the two measurement methods.

SECONDARY OUTCOMES:
Mean difference in diastolic blood pressure (mmHg) between guideline-based and routine clinical measurement | 1 year
  As above, for diastolic blood pressure (DBP).
Mean difference in mean arterial pressure (mmHg) between guideline-based and routine clinical measurement | 1 yaer
  Mean arterial pressure (MAP) will be calculated as MAP = (SBP + 2×DBP) / 3 for each measurement method. The outcome will be the within-participant difference between methods

CONTACTS AND LOCATIONS:
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel, Israel